CLINICAL TRIAL: NCT04267679
Title: Prospective Evaluation of Cannabidiol (CBD) on Anxiety: A Pilot Study
Brief Title: Cannabidiol for Anxiety
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped due to COVID-19 pandemic.
Sponsor: CB2 Insights (Other)
Collaborators: Green Lotus Hemp (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GL-2020
Record Dates: First submitted 2020-02-06; First posted 2020-02-13 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cannabidiol (Experimental): Participants will take 25 mg full-spectrum CBD soft gel capsules (2 to 4 per day) for 12 weeks.
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — 25 mg full-spectrum CBD soft gel capsules

SUMMARY:
This pilot trial seeks to investigate the effect of 25 mg full-spectrum CBD soft gel capsules (up to a total dosage of 100mg per day) on individuals with diagnosed anxiety. All participants will take CBD soft gel capsules for 12 weeks, and will be assessed at 6 weeks and 12 weeks post-enrollment using measures of anxiety, sleep and perception of change.

ELIGIBILITY:
1. Male or female patients 18 years of age or older with a GAD-7 score of 10 or greater
2. Presenting to a participating clinic for initial evaluation for a medical cannabis card
3. Willingness to abstain from the use of all other cannabis products for the trial period (3 months)
4. Not pregnant or planning to become pregnant during the trial period (3 months)
5. Not breastfeeding or planning to breastfeed during the trial period (3 months)
6. No history of cannabis use within 4 weeks of enrollment
7. No history of lifetime cannabis use disorder or other substance use disorders (except: tobacco use disorder)
8. No history of lifetime daily cannabis use
9. No family history of psychosis (e.g., bipolar disorder or schizophrenia)
10. No history of adverse reactions to cannabis
11. No recent changes to prescribed anxiety medications (within the last 1 month)
12. Provision of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder 7-item scale | 12 weeks
  The Generalized Anxiety Disorder 7-item scale is one of the most frequently used, validated self-reported questionnaires that is used to screen for, diagnose, and assess severity of generalized anxiety disorder.

SECONDARY OUTCOMES:
Perception of change | 12 weeks
  Participants will complete the Patients' Global Impression of Change (PGIC) scale at each follow-up visit, which has been regarded as an important self-reported indicator of change.
Protocol Compliance | 12 weeks
  Participants will self-report their intervention compliance using a simple log that will be provided to them at their enrollment visit and will be asked to bring their CBD log to every follow-up visit. Participants will also self-report any medical cannabis or opioid usage.
Sleep quality | 12 weeks
  Participants will be asked whether they believe that the CBD intervention has impacted their sleep quality. They will be asked to complete a short 2-question survey.